CLINICAL TRIAL: NCT06430203
Title: Indigenous Youth and Young Adults With Diabetes Peer Mentorship Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Romina Pace, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10728
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Distress, Emotional
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-mentoring (Experimental): Peer-mentoring which will include land based activities, nutrition and physical activity teaching.
  Interventions: Behavioral: Peer mentoring

INTERVENTIONS:
Behavioral: Peer mentoring — Indigenous young adult peer mentors who will develop and deliver the program based on needs and wants of our participants. The program will be built on their experience and ideas. They will be empowered to guide the program in the direction they see best for their communities.

SUMMARY:
The goal of this study is to learn if an Indigenous led peer-mentor program can provide Indigenous youth and young adults with the support needed to improve their distress and improve their diabetes control. Also, we will learn about Indigenous youth and young adults experience with diabetes.

* Can a peer-mentoring program reduce diabetes distress among Indigenous youth and young adults with diabetes?
* What is it like for Indigenous youth and young adults to be live with diabetes?
* Can a peer-mentoring program reduce global distress and improve resilience among Indigenous youth and young adults with diabetes?
* Can a peer-mentoring program lead to changes in lifestyle (diet, physical activity, substance use) and diabetes related clinical outcomes among Indigenous youth and young adults with diabetes.

Researchers will compare distress, resilience, lifestyles, and diabetes related clinical outcomes before participating in the peer-mentoring program and at 6 and 12 months into the program. Additionally, participants will be asked to share their journey with diabetes through photos throughout the program

Participants will:

* Be paired with peer-mentors who also have diabetes and they will share their journey with diabetes
* Participate in activities (grocery tours, walking clubs, land-based activities, cooking classes) held by peer-mentors
* Complete questionnaires on distress, resilience, and lifestyle every 6 months.
* Participate in Photovoice workshops to share their stories through pictures.

DETAILED DESCRIPTION:
The rates of diabetes are increasing among youth and young adults. This rise is particularly steep among Indigenous peoples who also face high rates of depression and emotional distress due to the ongoing legacy of colonization resulting in systemic racism and intergenerational trauma. Diabetes care includes many aspects of self-care (checking sugar, taking medication, following exercise and diet advice), which is negatively impacted by emotional distress. The emotional distress specific to living with diabetes, known as diabetes distress (DD), is due to feeling overwhelmed by the demands of self-care, fears of complications, and guilt or shame over lifestyle choices. DD is known to be related to decreased wellbeing and poor diabetes control. The rate of DD has not been studied among Indigenous youth, nor have interventions aimed at reducing it to improve diabetes management.

Peer support has been shown to help empower youth and young adults by normalizing their experiences and providing a safe space to express themselves. In the Eeyou Istchee Cree community in Quebec, Jonathan Linton, an Indigenous young adult with diabetes, developed a program for youth with diabetes on management and self-care for diabetes that incorporates traditional elements. As he helps participants be more active and eat healthier, he supports them in their journey with diabetes and creates a safe space for them to voice concerns, easing their distress.

This research study will build on the initiative developed by Mr. Linton to create a community of peer-mentors to provide Indigenous youth and young adults with the support needed to improve their distress and improve their diabetes control. To evaluate the program, a combination of questionnaires to assess changes in DD and other emotional factors, measures of diabetes outcomes (glycemia, blood pressure, weight), and Photovoice, a research tool that allows participants to use images to explain their experience with diabetes, will be used.

ELIGIBILITY:
Inclusion Criteria:

Age 10-29 years old Clinical diagnosis of diabetes or gestational diabetes

Exclusion Criteria:

Age > 29 years old Not at risk of diabetes

Ages: 10 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | 0,6 and 12 months
  Problem Areas in Diabetes (PAID) scale from 0-100, higher score means more distress

SECONDARY OUTCOMES:
Global Distress | 0,6 and 12 months
  0 item Kessler Psychological Distress scale (K10), from 10-50, the higher the score the greater the global distress.
Resilience-Children | 0,6 and 12 months
  Child and Youth Resilience Measure-Revised (CYRM-R), for 10-18 years old. Scale from 17-85, the higher the score the greater the resilience
Resilience-Adults | 0,6 and 12 months
  Adult Resilience Measure-Revised (ARM-R), for those > 18 years. Scale from 17-85, the higher the score the greater the resilience
Body Mass Index | 0 and 12 months
  Weight (kg)/[Height(m)]^2
Hemoglobin A1c | 0 and 12 months
  Percent HbA1c
urine albumin to creatine ratio | 0 and 12 months
  mg/mmol
low density lipoprotein | 0 and 12 months
  mmol/L
Blood pressure | 0 and 12 months
  mmHg
Lifestyle questionnaire | 0 and 12 months
  Developed by Cree Board of health to assess diet and physical activity. Not a scale

CONTACTS AND LOCATIONS:
Overall Officials: Romina Pace, Principal Investigator — MUHC-RI

IPD SHARING:
Plan to Share IPD: No